CLINICAL TRIAL: NCT01132274
Title: Near Zero Fluoroscopic Exposure During Catheter Ablation of Supraventricular Arrhythmias
Brief Title: Radiation Exposure Reduction in Supraventricular Tachycardia Ablation
Acronym: NO-PARTY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Abbott Medical Devices (Industry); CNR Institute of Clinical Physiology, Pisa, Italy (Unknown)
Responsible Party: Michela Casella, MD, PhD, Cardiac Arrhythmia Research Centre, Department of Cardiovascular Medicine, Centro Cardiologico Monzino, University of Milan, Milan, Italy
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSC210210
Record Dates: First submitted 2010-03-04; First posted 2010-05-28 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Supraventricular Tachycardias
Keywords: Supraventricular arrhythmia catheter ablation
MeSH Terms: conditions — Tachycardia, Supraventricular | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional catheter ablation (Active Comparator): Radiofrequency catheter ablation through fluoroscopic guidance
  Interventions: Procedure: Radiofrequency catheter ablation
- Non-fluoroscopic catheter ablation (Experimental): Radiofrequency catheter ablation guided by the EnSite NavX (St.Jude Medical, St Paul, MN, USA) mapping-system
  Interventions: Procedure: Radiofrequency catheter ablation

INTERVENTIONS:
Procedure: Radiofrequency catheter ablation — Conventional radiofrequency catheter ablation through fluoroscopic guidance of supraventricular arrhythmias.
  Arms: Conventional catheter ablation
Procedure: Radiofrequency catheter ablation — Radiofrequency catheter ablation through the non-fluoroscopic EnSite NavX mapping system (St.Jude Medical, St Paul, MN, USA) guidance.
  Arms: Non-fluoroscopic catheter ablation

SUMMARY:
Radiofrequency catheter ablation (RFCA) is the mainstay of therapy for supraventricular tachyarrhythmias, providing cure in a high percentage of cases. Conventional ablation techniques require the use of fluoroscopy to place and navigate catheters in the heart, thus exposing patients to ionizing radiations with an additional risk of cancer. The feasibility and safety of a non-fluoroscopic RFCA of a wide range of supraventricular arrhythmias using the EnSite NavX mapping system have been recently reported. The NO-PARTY is a multicenter, randomized-controlled trial designed to test the hypothesis that supraventricular arrhythmias RFCA through the non-fluoroscopic EnSite NavX mapping system results in a clinically significant reduction of the exposure to ionizing radiations compared with conventional ablation techniques.

NO-PARTY trial will determine whether supraventricular tachyarrhythmia RFCA through a non-fluoroscopic EnSite NavX mapping system is a suitable and cost-effective approach to achieve a clinically significant reduction of ionizing radiation exposure for both the patient and the operator.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients between 14 and 50 years of age who have received an indication to radiofrequency catheter ablation of supraventricular arrhythmias according to current guidelines.

Exclusion Criteria:

* atrial fibrillation or non isthmus-dependent atrial flutter
* pregnancy
* hematological contraindications to ionizing radiation exposure
* presence of complex congenital heart disease, and cardiac surgery within 1 month from enrollment

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Actual)
Dates: Start 2009-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
reduction of ionizing radiation exposure | 1 day (radiation exposure will be evaluated at the end of procedure)
  the NO-PARTY trial was designed to compare a non-fluoroscopic catheter ablation guided by the EnSite NavXTM mapping system with conventional catheter ablation for supraventricular tachyarrhythmias in terms of ionizing radiation exposure for both the patient and the operator

SECONDARY OUTCOMES:
Cost-Effectiveness | at 1 year
  The total reduction in fluoroscopy use with the non-fluoroscopic NavX mapping system approach is associated with a life-term ionizing radiation-exposure risk reduction, which will be estimated according to currently available ionizing radiation risk charts. Cost-effectiveness analysis will be performed taking into account such risk reduction, and the increased costs associated with the use of the nonfluoroscopic radiofrequency ablation approach.
Cost-Effectiveness | at 2 years
  The total reduction in fluoroscopy use with the non-fluoroscopic NavX mapping system approach is associated with a life-term ionizing radiation-exposure risk reduction, which will be estimated according to currently available ionizing radiation risk charts. Cost-effectiveness analysis will be performed taking into account such risk reduction, and the increased costs associated with the use of the nonfluoroscopic radiofrequency ablation approach.

CONTACTS AND LOCATIONS:
Overall Officials: Michela Casella, MD, PhD, Principal Investigator — Cardiac Arrhythmia Research Centre, Centro Cardiologico Monzino, University of Milan, Milan, Italy
Locations (6):
- Italy (6):
  - Santa Maria della Misericordia - A.O. di Perugia, Perugia, PG
  - Arrhythmia Department, Azienda Ospedaliero-Universitaria Pisana, Pisa, PI
  - CNR, Institute of Clinical Physiology, Fondazione G. Monasterio, Pisa, PI
  - Institute of Cardiology; Presidio Ospedaliero Santa Chiara, Trento, TN
  - Cardiac Arrhythmia Research Centre, Centro Cardiologico Monzino, University of Milan, Milan
  - Catholic University of the Sacred Heart, Rome

REFERENCES:
- [Background] Casella M, Dello Russo A, Pelargonio G, Bongiorni MG, Del Greco M, Piacenti M, Andreassi MG, Santangeli P, Bartoletti S, Moltrasio M, Fassini G, Marini M, Di Cori A, Di Biase L, Fiorentini C, Zecchi P, Natale A, Picano E, Tondo C. Rationale and design of the NO-PARTY trial: near-zero fluoroscopic exposure during catheter ablation of supraventricular arrhythmias in young patients. Cardiol Young. 2012 Oct;22(5):539-46. doi: 10.1017/S1047951112000042. Epub 2012 Feb 13. PMID 22325367
- [Derived] Casella M, Dello Russo A, Pelargonio G, Del Greco M, Zingarini G, Piacenti M, Di Cori A, Casula V, Marini M, Pizzamiglio F, Zucchetti M, Riva S, Russo E, Narducci ML, Soldati E, Panchetti L, Startari U, Bencardino G, Perna F, Santangeli P, Di Biase L, Cichocki F, Fattore G, Bongiorni M, Picano E, Natale A, Tondo C. Near zerO fluoroscopic exPosure during catheter ablAtion of supRavenTricular arrhYthmias: the NO-PARTY multicentre randomized trial. Europace. 2016 Oct;18(10):1565-1572. doi: 10.1093/europace/euv344. Epub 2015 Nov 10. PMID 26559916